CLINICAL TRIAL: NCT02394743
Title: Correlation Between Estimated Glomerular Filtration Rate(eGFR) and Vascular Inflammation Measured by Positron Emission Tomography (PET) With 18F-fluoro-deoxyglucose (FDG)
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Medical professor, Korea University
Other Study IDs: PET_eGRF
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Atherosclerosis
Keywords: Glomerular Filtration Rate
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- eGFR > 90: group whose eGFR is more than 90
  Interventions: Radiation: 18FDG-PET
- 60 < eGFR <90: group whose eGFR is between 60 and 90
  Interventions: Radiation: 18FDG-PET
- eGFR < 60: group whose eGFR is less than 60
  Interventions: Radiation: 18FDG-PET

INTERVENTIONS:
Radiation: 18FDG-PET

SUMMARY:
Vascular inflammation is a key factor in both the pathogenesis and outcome of atherosclerosis. Renal insufficiency is close correlation with atherosclerosis and cardiovascular mortality.

18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising tool for identifying and quantifying vascular inflammation within atherosclerotic plaques.Therefore, the purpose of the study is to demonstrate the correlation between eGFR and vascular inflammation detected by 18F FDG-PET.

ELIGIBILITY:
Inclusion Criteria:

1. absence of prior cancer diagnosis or remission from cancer at the time of PET imaging and throughout the follow-up period;
2. >=30 years of age;
3. no prior history of cardiovascular disease ; and
4. absence of acute or chronic inflammatory or autoimmune disease (based on documented medical history) or use of chronic anti-inflammatory therapy.

Exclusion Criteria:

1. age <35 years
2. presence of chronic inflammatory disease
3. use of anti-inflammatory medications
4. presence of active malignant cancer (defined as any radiological or pathological evidence of malignant cancer disease or undergoing chemotherapy or radiation therapy within 1 year before initial PET/CT and throughout the inter-scan duration).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who took 18FDG- PET in Korea Guro University
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2011-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Correlation between vascular inflammatory status measured by 18F FDG-PET and eGFR by Modification of Diet in Renal Disease(MDRD) formula | at 1 day of taking 18F FDG - PET

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Korea University College of Medicine, Seoul, VD, South Korea